CLINICAL TRIAL: NCT00069095
Title: A 2x2 Factorial Randomized Phase III Study of Intermittent Oral Capecitabine in Combination With Intravenous Oxaliplatin (Q3W) ("XELOX") With/Without Intravenous Bevacizumab (Q3W) Versus Bolus and Continuous Infusion Fluorouracil/Intravenous Leucovorin With Intravenous Oxaliplatin (Q2W) ("FOLFOX-4") With/Without Intravenous Bevacizumab (Q2W) as First-line Treatment for Patients With Metastatic Colorectal Cancer
Brief Title: A Study of Capecitabine (Xeloda) and Bevacizumab as a First-line Therapy in Patients With Metastatic Colorectal Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: NO16966
Record Dates: First submitted 2003-09-15; First posted 2003-09-18 (Estimated); Results first posted 2016-01-22 (Estimated); Last update posted 2016-10-06 (Estimated); Status verified 2016-08

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Oxaliplatin; Capecitabine; Bevacizumab; Leucovorin; Fluorouracil

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (4):
- XELOX (oxaliplatin+capecitabine) (Experimental): Patients in the 2-arm part of the study received oxaliplatin 130 mg/m^2 intravenously (iv) on Day 1 of every 3 week cycle + capecitabine 1000 mg/m^2 orally twice a day for the first 2 weeks of every 3 week cycle. Patients in the 4-arm part of the study received the same treatments plus placebo for bevacizumab 7.5 mg/kg iv on Day 1 of every 3 week cycle.
  Interventions: Drug: Oxaliplatin 130 mg/m^2; Drug: Capecitabine 1000 mg/m^2; Drug: Placebo for bevacizumab 7.5 mg/kg
- XELOX (oxaliplatin+capecitabine) + bevacizumab (Experimental): Patients in the 4-arm part of the study received oxaliplatin 130 mg/m^2 intravenously (iv) on Day 1 of every 3 week cycle + capecitabine 1000 mg/m^2 orally twice a day for the first 2 weeks of every 3 week cycle + bevacizumab 7.5 mg/kg iv on Day 1 of every 3 week cycle.
  Interventions: Drug: Oxaliplatin 130 mg/m^2; Drug: Capecitabine 1000 mg/m^2; Drug: Bevacizumab 7.5 mg/kg
- FOLFOX-4 (oxaliplatin+leucovorin+fluorouracil) (Active Comparator): Patients in the 2-arm part of the study received oxaliplatin 85 mg/m^2 intravenously (iv) + leucovorin 200 mg/m^2 iv on Day 1 of every 2 week cycle + fluorouracil 400 mg/m^2 bolus injection over 2 to 4 min followed by 600 mg/m^2 continuous infusion over 22 h on Days 1 and 2 of every 2 week cycle. Patients in the 4-arm part of the study received the same treatments plus placebo for bevacizumab 5 mg/kg iv on Day 1 of every 2 week cycle.
  Interventions: Drug: Oxaliplatin 85 mg/m^2; Drug: Leucovorin 200 mg/m^2; Drug: Fluorouracil 400 mg/m^2; Drug: Placebo for bevacizumab 5 mg/kg
- FOLFOX-4 (oxaliplatin+leucovorin+fluorouracil) + bevacizumab (Active Comparator): Patients in the 4-arm part of the study received oxaliplatin 85 mg/m^2 intravenously (iv) + leucovorin 200 mg/m^2 iv + bevacizumab 5 mg/kg iv on Day 1 of every 2 week cycle + fluorouracil 400 mg/m^2 bolus injection over 2 to 4 min followed by 600 mg/m^2 continuous infusion over 22 h on Days 1 and 2 of every 2 week cycle.
  Interventions: Drug: Oxaliplatin 85 mg/m^2; Drug: Leucovorin 200 mg/m^2; Drug: Fluorouracil 400 mg/m^2; Drug: Bevacizumab 5 mg/kg

INTERVENTIONS:
Drug: Oxaliplatin 130 mg/m^2 — Oxaliplatin was administered in a 2 h infusion before the first dose of capecitabine.
  Other Names: Eloxatin
  Arms: XELOX (oxaliplatin+capecitabine); XELOX (oxaliplatin+capecitabine) + bevacizumab
Drug: Capecitabine 1000 mg/m^2 — Capecitabine was taken within 30 min after the end of breakfast and dinner.
  Other Names: Xeloda
  Arms: XELOX (oxaliplatin+capecitabine); XELOX (oxaliplatin+capecitabine) + bevacizumab
Drug: Bevacizumab 7.5 mg/kg — Bevacizumab was administered in a 30 to 90 min infusion.
  Other Names: Avastin
  Arms: XELOX (oxaliplatin+capecitabine) + bevacizumab
Drug: Placebo for bevacizumab 7.5 mg/kg — Placebo control for bevacizumab (volume equivalent to 7.5 mg/kg bevacizumab) was administered in a 30 to 90 min infusion.
  Arms: XELOX (oxaliplatin+capecitabine)
Drug: Oxaliplatin 85 mg/m^2 — Oxaliplatin 85 mg/m^2 was administered simultaneously with leucovorin in a 2 h infusion.
  Other Names: Eloxatin
  Arms: FOLFOX-4 (oxaliplatin+leucovorin+fluorouracil); FOLFOX-4 (oxaliplatin+leucovorin+fluorouracil) + bevacizumab
Drug: Leucovorin 200 mg/m^2 — Leucovorin was administered simultaneously with oxaliplatin 85 mg/m^2 in a 2 h infusion.
  Arms: FOLFOX-4 (oxaliplatin+leucovorin+fluorouracil); FOLFOX-4 (oxaliplatin+leucovorin+fluorouracil) + bevacizumab
Drug: Fluorouracil 400 mg/m^2
  Other Names: Efudex
  Arms: FOLFOX-4 (oxaliplatin+leucovorin+fluorouracil); FOLFOX-4 (oxaliplatin+leucovorin+fluorouracil) + bevacizumab
Drug: Bevacizumab 5 mg/kg — Bevacizumab was administered in a 30 to 90 min infusion.
  Other Names: Avastin
  Arms: FOLFOX-4 (oxaliplatin+leucovorin+fluorouracil) + bevacizumab
Drug: Placebo for bevacizumab 5 mg/kg — Placebo control for bevacizumab (volume equivalent to 5 mg/kg bevacizumab) was administered in a 30 to 90 min infusion.
  Arms: FOLFOX-4 (oxaliplatin+leucovorin+fluorouracil)

SUMMARY:
This 4 arm study assessed the efficacy and safety of oral capecitabine (Xeloda) or intravenous (iv) fluorouracil/leucovorin, in combination with iv oxaliplatin (Eloxatin) with or without iv bevacizumab (Avastin), as a first-line treatment in patients with metastatic colorectal cancer. Patients were randomized to receive 1) XELOX (Xeloda 1000 mg/m^2 orally [po] twice a day [bid] on Days 1-15 + oxaliplatin in 3 week cycles), 2) FOLFOX-4 (oxaliplatin + leucovorin + fluorouracil [5-FU] in 2 week cycles), 3) XELOX + bevacizumab (7.5 mg iv on Day 1 in 3 week cycles), or 4) FOLFOX-4 + bevacizumab (5 mg iv on Day 1 in 2 week cycles).

DETAILED DESCRIPTION:
This study was conducted in 2 parts: An initial 2-arm part in which patients were randomized to 1 of 2 different treatment groups (XELOX or FOLFOX-4), and a subsequent 2 x 2 factorial part, added to the study through a protocol amendment, in which additional patients were randomized into one of 4 different treatment groups (XELOX + placebo, FOLFOX-4 + placebo, XELOX + bevacizumab, or FOLFOX-4 + bevacizumab). Due to the comparison of the oral agent capecitabine with bolus and infused fluorouracil, the study was not blinded with respect to these 2 treatments. The study was double-blind with regard to the administration of bevacizumab, ie, there was a placebo control for bevacizumab in the second part of the study.

The study consisted of 3 phases, a Primary Study Treatment Phase, a Post-Study Treatment Phase, and a Follow-Up Phase.

Primary Study Treatment Phase

Patients were to receive up to 16 cycles (2-arm part of the study) or 24 cycles (4-arm part of the study) of treatment during the Primary Study Treatment Phase (48 weeks).

Post-Study Treatment Phase

Patients who completed the 48-week primary study treatment phase without progressive disease were eligible to enter the post-study treatment phase at the discretion of the investigator and the sponsor. Patients who entered this phase were to continue treatment on the same regimen to which they were initially randomized until either progression of disease was documented, unacceptable toxicity occurred, or the patient withdrew consent.

Follow-up Phase

Patients who terminated study treatment during the primary or post-study treatment phase were followed until disease progression or death.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients ≥ 18 years of age.
* Metastatic colorectal cancer.
* ≥ 1 target lesion.

Exclusion Criteria:

* Previous treatment with oxaliplatin or bevacizumab.
* Previous systemic chemotherapy or immunotherapy for advanced or metastatic disease.
* Progressive disease during or within 6 months of completion of previous adjuvant therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2035 (Actual)
Dates: Start 2003-07; Primary Completion 2006-01 (Actual); Study Completion 2009-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (205):
- United States (47):
  - Berkeley, California
  - Fountain Valley, California
  - Fullerton, California
  - Gilroy, California
  - Greenbrae, California
  - Los Angeles, California
  - Orange, California
  - Palo Alto, California
  - San Diego, California
  - Norwich, Connecticut
  - Waterbury, Connecticut
  - Boca Raton, Florida
  - Gainesville, Florida
  - Jacksonville, Florida
  - New Port Richey, Florida
  - Tampa, Florida
  - Atlanta, Georgia
  - Chicago, Illinois
  - Elk Grove Village, Illinois
  - Peoria, Illinois
  - Lexington, Kentucky
  - New Orleans, Louisiana
  - Scarborough, Maine
  - Boston, Massachusetts
  - Ann Arbor, Michigan
  - Saint Louis Park, Minnesota
  - Las Vegas, Nevada
  - East Orange, New Jersey
  - Hamilton, New Jersey
  - New Brunswick, New Jersey
  - Albuquerque, New Mexico
  - Farmington, New Mexico
  - New York, New York
  - Rochester, New York
  - Syracuse, New York
  - Charlotte, North Carolina
  - Bismarck, North Dakota
  - Fargo, North Dakota
  - Sayre, Pennsylvania
  - Upland, Pennsylvania
  - Providence, Rhode Island
  - Charleston, South Carolina
  - Columbia, South Carolina
  - Memphis, Tennessee
  - Houston, Texas
  - Burlington, Vermont
  - Richmond, Virginia
- Australia (13):
  - Adelaide
  - Box Hill
  - Brisbane
  - Camperdown
  - Fitzroy
  - Footscray
  - Kurralta Park
  - Malvern
  - Melbourne
  - Perth
  - Port Macquarie
  - St Leonards
  - Sydney
- Austria (2):
  - Vienna
  - Wels
- Brazil (3):
  - Jaú
  - Rio de Janeiro
  - São Paulo
- Canada (19):
  - Calgary, Alberta
  - Edmonton, Alberta
  - Kelowna, British Columbia
  - North Vancouver, British Columbia
  - Surrey, British Columbia
  - Vancouver, British Columbia
  - Victoria, British Columbia
  - Winnipeg, Manitoba
  - Halifax, Nova Scotia
  - Hamilton, Ontario
  - London, Ontario
  - Mississauga, Ontario
  - Oshawa, Ontario
  - Ottawa, Ontario
  - St. Catharines, Ontario
  - Toronto, Ontario
  - Lévis, Quebec
  - Montreal, Quebec
  - Québec, Quebec
- China (9):
  - Beijing
  - Guangdong
  - Guangzhou
  - Jiangsu
  - Jiangxi
  - Shandong
  - Shanghai
  - Tianjin
  - Wuhan
- Czechia (4):
  - Brno
  - Chomutov
  - Hradec Králové
  - Ostrava
- Denmark (3):
  - Copenhagen
  - Herlev
  - Odense
- Finland (3):
  - Helsinki
  - Tampere
  - Turku
- France (17):
  - Besançon
  - Bobigny
  - Boulogne-Billancourt
  - Brest
  - Chambray-lès-Tours
  - Colmar
  - Dijon
  - Grenoble
  - Lyon
  - Metz
  - Nice
  - Nîmes
  - Paris
  - Pierre-Bénite
  - Rouen
  - Saint-Herblain
  - Toulouse
- Germany (10):
  - Bochum
  - Halle
  - Hanover
  - Herne
  - Leipzig
  - Mainz
  - Mannheim
  - Regensburg
  - Stralsund
  - Trier
- Guatemala City, Guatemala
- Hong Kong, Hong Kong
- Hungary (3):
  - Budapest
  - Győr
  - Kecskemét
- Ireland (3):
  - Cork
  - Dublin
  - Galway
- Israel (5):
  - Haifa
  - Jerusalem
  - Petah Tikva
  - Tel Aviv
  - Ẕerifin
- Italy (8):
  - Ancona
  - Genova
  - Modena
  - Padua
  - Parma
  - Pavia
  - Reggio Emilia
  - Sassari
- Mexico City, Mexico
- Christchurch, New Zealand
- Norway (3):
  - Bergen
  - Oslo
  - Tromsø
- Panama City, Panama
- Portugal (2):
  - Beja
  - Lisbon
- San Juan, Puerto Rico
- Russia (2):
  - Moscow
  - Saint Petersburg
- South Africa (3):
  - Cape Town
  - Pretoria
  - Sandton
- Seoul, South Korea
- Spain (9):
  - Barcelona
  - Córdoba
  - Granada
  - Leganés
  - Madrid
  - Málaga
  - Santander
  - Valencia
  - Zaragoza
- Sweden (5):
  - Gävle
  - Karlstad
  - Stockholm
  - Uppsala
  - Västerås
- Switzerland (2):
  - Bern
  - Geneva
- Taiwan (2):
  - Kueishan
  - Taipei
- Thailand (2):
  - Bangkok
  - Khon Kaen
- Turkey (Türkiye) (2):
  - Istanbul
  - Izmir
- United Kingdom (17):
  - Aberdeen
  - Birmingham
  - Cardiff
  - Derby
  - Glasgow
  - Guildford
  - Hull
  - London
  - Maidstone
  - Newcastle upon Tyne
  - Northwood
  - Nottingham
  - Plymouth
  - Salisbury
  - Southampton
  - Sutton
  - Taunton

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted in 32 countries - Australia, Austria, Brazil, Canada, China, Czech Republic, Denmark, Finland, France, Germany, Great Britain, Guatemala, Hong Kong, Hungary, Ireland, Israel, Italy, Korea, Mexico, New Zealand, Norway, Panama, Portugal, Russia, South Africa, Spain, Sweden, Switzerland, Taiwan, Thailand, Turkey and USA.
Pre-assignment Details: A total of 2035 participants were randomized to any one of the treatment groups in the study (634 participants in the initial 2-arm part and 1401 participants in the 2x2 factorial part of the study), but only 2034 received study treatment as 1 participant was enrolled twice in the study at 2 study centers.
Groups:
- Xelox: Participants in the 2-arm part of the study received intravenous infusion of oxaliplatin 130 mg/m^2 over 2 hours on Day 1 of every 3 weeks before the first dose of capecitabine. Capecitabine was administered orally within 30 minutes after the end of a meal (breakfast and dinner) at a dose of 1000 mg/m^2 twice-daily (equivalent to a total daily dose of 2000 mg/m^2), for the first 2 weeks of every 3-week cycle. Participants received up to 16 cycles of treatment during the primary study treatment phase (48 weeks). Participants who completed the 48-week primary study treatment phase without progressive disease were eligible to enter the post-study treatment phase at the discretion of the investigator and the sponsor. Participants who entered this phase were to continue treatment on the same regimen to which they were initially randomized until either progression of disease was documented, unacceptable toxicity occurred, or the participant withdrew consent.
- Folfox-4: Participants in the 2-arm part of the study received intravenous infusion of oxaliplatin 85 mg/m^2 on Day 1 of every 2-week cycle; concomitantly with leucovorin 200 mg/m^2 iv for 2 hours followed by fluorouracil 400 mg/m^2 bolus injection over 2 to 4 min followed by 600 mg/m^2 continuous infusion over 22 h on Days 1 and 2 of every 2-week cycle. Participants received up to 24 cycles of treatment during the primary study treatment phase (48 weeks). Participants who completed the 48-week primary study treatment phase without progressive disease were eligible to enter the post-study treatment phase at the discretion of the investigator and the sponsor. Participants who entered this phase were to continue treatment on the same regimen to which they were initially randomized until either progression of disease was documented, unacceptable toxicity occurred, or the participant withdrew consent.
- Xelox+P: Participants in the 2x2 factorial part of the study received intravenous infusion of placebo control for bevacizumab (BV) [volume equivalent to 7.5 mg/kg BV] over 30 to 90 minutes followed by oxaliplatin 130 mg/m^2 over 2 hours on Day 1 of every 3 weeks in combination with capecitabine, administered orally at a dose of 1000 mg/m^2 twice-daily (equivalent to a total daily dose of 2000 mg/m^2), for the first 2 weeks of every 3-week cycle. Participants received up to 16 cycles of treatment during the primary study treatment phase (48 weeks). Participants who completed the 48-week primary study treatment phase without progressive disease were eligible to enter the post-study treatment phase at the discretion of the investigator and the sponsor. Participants who entered this phase were to continue treatment on the same regimen to which they were initially randomized until either progression of disease was documented, unacceptable toxicity occurred, or the participant withdrew consent.
- Folfox-4+P: Participants in the 2x2 factorial part of the study received intravenous infusion of placebo control for BV (volume equivalent to 5 mg/kg BV) over 30 to 90 minutes followed by oxaliplatin 85 mg/m^2 on Day 1 of every 2-week cycle; concomitantly with leucovorin 200 mg/m^2 iv for 2 hours followed by fluorouracil 400 mg/m^2 bolus injection over 2 to 4 min followed by 600 mg/m^2 continuous infusion over 22 h on Days 1 and 2 of every 2-week cycle. Participants received up to 24 cycles of treatment during the primary study treatment phase (48 weeks). Participants who completed the 48-week primary study treatment phase without progressive disease were eligible to enter the post-study treatment phase at the discretion of the investigator and the sponsor. Participants who entered this phase were to continue treatment on the same regimen to which they were initially randomized until either progression of disease was documented, unacceptable toxicity occurred, or the participant withdrew consent.
- Xelox+BV: Participants in the 2x2 factorial part of the study received intravenous infusion of bevacizumab 7.5 mg/kg over 30 to 90 minutes followed by oxaliplatin 130 mg/m^2 over 2 hours on Day 1 of every 3 weeks in combination with capecitabine, administered orally at a dose of 1000 mg/m^2 twice-daily (equivalent to a total daily dose of 2000 mg/m^2), for the first 2 weeks of every 3-week cycle. Participants received up to 16 cycles of treatment during the primary study treatment phase (48 weeks). Participants who completed the 48-week primary study treatment phase without progressive disease were eligible to enter the post-study treatment phase at the discretion of the investigator and the sponsor. Participants who entered this phase were to continue treatment on the same regimen to which they were initially randomized until either progression of disease was documented, unacceptable toxicity occurred, or the participant withdrew consent.
- Folfox-4+BV: Participants in the 2x2 factorial part of the study received intravenous infusion of bevacizumab 5 mg/kg over 30 to 90 minutes followed by oxaliplatin 85 mg/m^2 on Day 1 of every 2-week cycle; concomitantly with leucovorin 200 mg/m^2 iv for 2 hours followed by fluorouracil 400 mg/m^2 bolus injection over 2 to 4 min followed by 600 mg/m^2 continuous infusion over 22 h on Days 1 and 2 of every 2-week cycle. Participants received up to 24 cycles of treatment during the primary study treatment phase (48 weeks). Participants who completed the 48-week primary study treatment phase without progressive disease were eligible to enter the post-study treatment phase at the discretion of the investigator and the sponsor. Participants who entered this phase were to continue treatment on the same regimen to which they were initially randomized until either progression of disease was documented, unacceptable toxicity occurred, or the participant withdrew consent.
Period: Primary Treatment Phase
Arm/Group | Xelox | Folfox-4 | Xelox+P | Folfox-4+P | Xelox+BV | Folfox-4+BV
Started | 317 | 317 | 350 | 351 | 350 | 349
Completed | 22 | 15 | 36 | 31 | 48 | 48
Not Completed | 295 | 302 | 314 | 320 | 302 | 301
Not completed — Ongoing | 0 | 0 | 5 | 7 | 7 | 4
Not completed — Admin/Other | 29 | 38 | 31 | 45 | 48 | 42
Not completed — Adverse Event | 99 | 92 | 71 | 72 | 109 | 101
Not completed — Death | 14 | 8 | 2 | 5 | 8 | 8
Not completed — Failure to return | 5 | 5 | 0 | 0 | 0 | 2
Not completed — Insufficient Therapeutic Response | 131 | 127 | 175 | 154 | 101 | 102
Not completed — Refused treatment | 15 | 26 | 17 | 31 | 24 | 27
Not completed — Withdrew | 2 | 3 | 8 | 2 | 4 | 9
Not completed — Other Violation | 0 | 1 | 1 | 1 | 0 | 1
Not completed — Violation criteria | 0 | 2 | 4 | 3 | 1 | 5
Period: Post-study Treatment Phase
Arm/Group | Xelox | Folfox-4 | Xelox+P | Folfox-4+P | Xelox+BV | Folfox-4+BV
Started | 8 (Participants could enter the follow-up phase even without entering the post-study treatment phase.) | 13 (Participants could enter the follow-up phase even without entering the post-study treatment phase.) | 21 (Participants could enter the follow-up phase even without entering the post-study treatment phase.) | 17 (Participants could enter the follow-up phase even without entering the post-study treatment phase.) | 36 (Participants could enter the follow-up phase even without entering the post-study treatment phase.) | 29 (Participants could enter the follow-up phase even without entering the post-study treatment phase.)
Completed | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 8 | 13 | 21 | 17 | 36 | 29
Not completed — Missing reason | 1 | 3 | 12 | 8 | 18 | 17
Not completed — Adverse Event | 2 | 3 | 1 | 0 | 5 | 1
Not completed — Eligible for surgery | 2 | 0 | 0 | 0 | 0 | 0
Not completed — Insufficient therapeutic response | 1 | 4 | 5 | 6 | 7 | 9
Not completed — Participant refusal/Admin reasons | 1 | 0 | 0 | 0 | 0 | 1
Not completed — Participant had complete response | 1 | 1 | 0 | 0 | 0 | 0
Not completed — More than 21 days delay between cycles | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Investigator decision (enough treatment) | 0 | 1 | 1 | 0 | 1 | 0
Not completed — Participant withdrew consent | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Participant will start new treatment | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Participant wanted break from treatment | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Participant completed treatment | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Surgery | 0 | 0 | 0 | 1 | 1 | 0
Not completed — Death | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Participant had progressive disease | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Participant/Physician decision to stop | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Preplanned 6 cycles after surgery | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Investigator decision | 0 | 0 | 0 | 0 | 0 | 1
Period: Follow-up Phase
Arm/Group | Xelox | Folfox-4 | Xelox+P | Folfox-4+P | Xelox+BV | Folfox-4+BV
Started | 284 (Participants could enter the follow-up phase even without entering the post-study treatment phase.) | 299 (Participants could enter the follow-up phase even without entering the post-study treatment phase.) | 298 (Participants could enter the follow-up phase even without entering the post-study treatment phase.) | 299 (Participants could enter the follow-up phase even without entering the post-study treatment phase.) | 278 (Participants could enter the follow-up phase even without entering the post-study treatment phase.) | 272 (Participants could enter the follow-up phase even without entering the post-study treatment phase.)
Completed | 110 | 93 | 178 | 187 | 186 | 171
Not Completed | 174 | 206 | 120 | 112 | 92 | 101
Not completed — Death | 174 | 206 | 120 | 112 | 92 | 101

BASELINE CHARACTERISTICS:
Population: Baseline characteristics were described for the Intent-to-treat (ITT) population.This population included all randomized participants who provided written informed consent.
Groups:
- Total: Total of all reporting groups
Arm/Group | Xelox | Folfox-4 | Xelox+P | Folfox-4+P | Xelox+BV | Folfox-4+BV | Total
Number analyzed (Participants) | 317 | 317 | 350 | 351 | 350 | 349 | 2034
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.3 (10.76) | 60.6 (10.94) | 59.1 (12.14) | 58.8 (10.87) | 59.7 (11.28) | 59.7 (10.74) | 59.7 (11.14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 123 | 113 | 145 | 165 | 137 | 144 | 827
  Male | 194 | 204 | 205 | 186 | 213 | 205 | 1207

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS) as Assessed by the Investigator According to Response Evaluation Criteria in Solid Tumors (RECIST) by General Approach (Participants With Curative Surgery Censored): Non-inferiority of XELOX Versus FOLFOX-4
Description: PFS was defined as the time from randomization to progressive disease or death. Participants with neither disease progression nor death were censored at the last date of the last tumor assessment that confirmed that their disease had not progressed. Participants with no tumor assessments after baseline who were alive at the time of clinical cutoff were censored at the date of randomization. Participants who underwent surgical resection with curative intent without prior progression were censored at the date of surgery. PFS was based on tumor assessments made by the investigators according to the RECIST criteria. Non-inferiority analysis that followed the general approach took into account all tumor assessments obtained during the primary study treatment phase, the post-study treatment phase and those obtained during the follow-up phase. Non-inferiority of the XELOX-containing arms compared with the FOLFOX-4- containing arms was investigated.
Time Frame: Baseline until disease progression or death, approximately 2 years 6 months
Population: The eligible patient population (EPP) excluded participants from the ITT who had violated major protocol inclusion or exclusion criteria or participants who were randomized and did not receive at least one dose of capecitabine, 5-FU, oxaliplatin, or bevacizumab/placebo.
Measure: Median (95% Confidence Interval); unit: days
Groups:
- FOLFOX-4/FOLFOX-4+P/FOLFOX-4+BV: Participants from the initial 2-arm part and the 2x2 factorial part of the study including the following groups -
  1. Folfox-4: Participants who received 2-week cycles of infused leucovorin, bolus injection fluorouracil and continuous infusion fluorouracil (given on days 1 and 2), combined with intravenous oxaliplatin (given on day 1).
  2. Folfox-4+P: Participants who received 2-week cycles of infused leucovorin, bolus injection fluorouracil and continuous infusion fluorouracil (given on days 1 and 2), combined with intravenous oxaliplatin and placebo control for bevacizumab (both given on day 1 every 2 weeks).
  3. Folfox-4+BV: Participants who received 2-week cycles of infused leucovorin, bolus injection fluorouracil and continuous infusion fluorouracil (given on days 1 and 2), combined with intravenous oxaliplatin and intravenous bevacizumab (both given on day 1 every 2 weeks).
- XELOX/XELOX+P/XELOX+BV: Participants from the initial 2-arm part and the 2x2 factorial part of the study including the following groups -
  1. Xelox: Capecitabine was administered as an oral twice-daily outpatient intermittent treatment (3-week cycles consisting of 2 weeks of treatment followed by 1 week without treatment) combined with intravenous oxaliplatin (given on day 1).
  2. Xelox+P: Capecitabine was administered as an oral twice-daily outpatient intermittent treatment (3-week cycles consisting of 2 weeks of treatment followed by 1 week without treatment) combined with intravenous oxaliplatin and placebo (P) control for bevacizumab (both given on day 1 every 3 weeks).
  3. Xelox+BV: Capecitabine was administered as an oral twice-daily outpatient intermittent treatment (3-week cycles consisting of 2 weeks of treatment followed by 1 week without treatment) combined with intravenous oxaliplatin and intravenous bevacizumab (both given on day 1 every 3 weeks).
Arm/Group | FOLFOX-4/FOLFOX-4+P/FOLFOX-4+BV | XELOX/XELOX+P/XELOX+BV
Number analyzed (Participants) | 937 | 967
days | 259 [245 to 268] | 241 [229 to 254]
Statistical Analysis 1: Comparison: FOLFOX-4/FOLFOX-4+P/FOLFOX-4+BV vs XELOX/XELOX+P/XELOX+BV; Equivalence of treatment arm A ('XELOX') to treatment arm B ('FOLFOX-4') was tested via the following hypotheses - H0: HRA/B >/= 1.23 versus H1: HRA/B < 1.23. HRA/B denotes the hazard of disease progression or death under treatment A ('XELOX') divided by the hazard of disease progression or death under treatment B ('FOLFOX-4'); Test type: Non-Inferiority or Equivalence — Non-inferiority was demonstrated if the upper limit of the 2-sided 97.5% confidence interval (CI) for the hazard ratio (HR) was less than the predefined limit of 1.23 (the non-inferiority margin). A stratified Cox model was used. In order to retain an experiment-wise two-sided type I error of 5%, the non-inferiority analysis for PFS used a two-sided significance level of 2.5%; Hazard Ratio (HR) = 1.05, 97.5% CI 2-sided [0.94 to 1.18]

2. Secondary Outcome: PFS as Assessed by the Independent Review Committee (IRC) (General Approach, Participants With Curative Surgery Censored) - Non-inferiority of XELOX Versus FOLFOX-4
Description: PFS is defined as the time from randomization to disease progression (PD) or death due to any cause. Participants with neither disease progression nor death were censored at the last date of the last tumor assessment that confirmed that their disease had not progressed. Participants who underwent surgical resection with curative intent without prior progression were censored at the date of surgery. PFS was analyzed on the basis of the tumor response assessments made by the IRC. Non-inferiority analysis that followed the general approach took into account all tumor assessments obtained during the primary study treatment phase, the post-study treatment phase and those obtained during the follow-up phase. Non-inferiority of the XELOX-containing arms was compared with the FOLFOX-4-containing arms.
Time Frame: Baseline until disease progression or death, approximately 2 years 6 months
Population: The EPP excluded participants from the ITT who had violated major protocol inclusion or exclusion criteria or participants who were randomized and did not receive at least one dose of capecitabine, 5-FU, oxaliplatin, or bevacizumab/placebo.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | FOLFOX-4/FOLFOX-4+P/FOLFOX-4+BV | XELOX/XELOX+P/XELOX+BV
Number analyzed (Participants) | 937 | 967
days | 304.0 [281 to 319] | 261.0 [246 to 276]
Statistical Analysis 1: Comparison: FOLFOX-4/FOLFOX-4+P/FOLFOX-4+BV vs XELOX/XELOX+P/XELOX+BV; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Hazard Ratio (HR) = 1.22, 97.5% CI 2-sided [1.05 to 1.42]

3. Secondary Outcome: PFS as Assessed by the Independent Review Committee (IRC) (General Approach, Participants With Curative Surgery Censored) - Superiority of Chemotherapy Plus BV Over Chemotherapy Alone
Description: PFS is defined as the time from randomization to disease progression (PD) or death due to any cause. Participants with neither disease progression nor death were censored at the last date of the last tumor assessment that confirmed that their disease had not progressed. Participants who underwent surgical resection with curative intent without prior progression were censored at the date of surgery. PFS was analyzed on the basis of the tumor response assessments made by the IRC. Superiority analysis that followed the general approach took into account all tumor assessments obtained during the primary study treatment phase, the post-study treatment phase and those obtained during the follow-up phase. Superiority of the bevacizumab-containing arms was compared with the placebo-containing arms.
Time Frame: Baseline until disease progression or death, approximately 2 years 6 months
Population: The ITT population included all randomized participants who provided written informed consent.
Measure: Median (95% Confidence Interval); unit: days
Groups:
- FOLFOX-4+P/XELOX+P: Participants from the 2x2 factorial part of the study including the following groups -
  1. Folfox-4+P: Participants received 2-week cycles of infused leucovorin, bolus injection fluorouracil and continuous infusion fluorouracil (given on days 1 and 2), combined with intravenous oxaliplatin and placebo control for bevacizumab (both given on day 1 every 2 weeks).
  2. Xelox+P: Capecitabine was administered as an oral twice-daily outpatient intermittent treatment (3-week cycles consisting of 2 weeks of treatment followed by 1 week without treatment) combined with intravenous oxaliplatin and placebo (P) control for bevacizumab (both given on day 1 every 3 weeks).
- FOLFOX-4+BV/XELOX+BV: Participants from the 2x2 factorial part of the study including the following groups -
  1. Folfox-4+BV: Participants who received 2-week cycles of infused leucovorin, bolus injection fluorouracil and continuous infusion fluorouracil (given on days 1 and 2), combined with intravenous oxaliplatin and intravenous bevacizumab (both given on day 1 every 2 weeks).
  2. Xelox+BV: Capecitabine was administered as an oral twice-daily outpatient intermittent treatment (3-week cycles consisting of 2 weeks of treatment followed by 1 week without treatment) combined with intravenous oxaliplatin and intravenous bevacizumab (both given on day 1 every 3 weeks).
Arm/Group | FOLFOX-4+P/XELOX+P | FOLFOX-4+BV/XELOX+BV
Number analyzed (Participants) | 701 | 699
days | 259.0 [244 to 278] | 335.0 [310 to 363]
Statistical Analysis 1: Comparison: FOLFOX-4+P/XELOX+P vs FOLFOX-4+BV/XELOX+BV; Testing for superiority was based on the stratified log-rank test and used a two-sided significance level of 2.5%.The hazard ratio (HR) of bevacizumab in combination with chemotherapy versus chemotherapy alone [HR(FOLFOX-4+P/XELOX+P)/(FOLFOX-4+BV/XELOX+BV)] was presented; Test type: Superiority or Other; p < 0.0001, Log Rank; Hazard Ratio (HR) = 0.70, 97.5% CI 2-sided [0.58 to 0.83]

4. Secondary Outcome: PFS (On-treatment Approach): Non-inferiority of XELOX Versus FOLFOX-4
Description: PFS is defined as the time from randomization to disease progression (PD) or death due to any cause. The on-treatment analysis included only tumor assessments and death events that occurred no later than 28 days after the last confirmed intake of any study medication in the primary study treatment phase. Participants who did not have an event during this interval were censored at the date of the last tumor assessment within this time window, or on day 1 if no tumor assessment was available after baseline. Participants who underwent surgical resection with curative intent without prior progression within 28 days after the last confirmed intake of any study medication in the primary study treatment phase were censored at the date of surgery. The on-treatment approach excluded the possible impact of other treatments that might have been started before disease progression. Non-inferiority of the XELOX-containing arms was compared with the FOLFOX-4-containing arms.
Time Frame: Baseline until disease progression or death, approximately 2 years 6 months
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | FOLFOX-4/FOLFOX-4+P/FOLFOX-4+BV | XELOX/XELOX+P/XELOX+BV
Number analyzed (Participants) | 937 | 967
days | 268.0 [252 to 290] | 234.0 [221 to 251]
Statistical Analysis 1: Comparison: FOLFOX-4/FOLFOX-4+P/FOLFOX-4+BV vs XELOX/XELOX+P/XELOX+BV; HRs and 97.5% confidence interval were reported for treatment arm A (XELOX/XELOX+P/XELOX+BV) versus treatment arm B (FOLFOX-4/FOLFOX-4+P/FOLFOX-4+BV); Test type: Non-Inferiority or Equivalence — Fewer events were expected in the 'on-treatment analysis', thus leading to reduced power. No formal statistical testing was therefore applied; Hazard Ratio (HR) = 1.24, 97.5% CI 2-sided [1.07 to 1.44]

5. Secondary Outcome: PFS (On-treatment Approach): Superiority of Chemotherapy Plus BV Over Chemotherapy Alone
Description: as for outcome 4
Time Frame: Baseline until disease progression or death, approximately 2 years 6 months
Population: The ITT population included all randomized participants who provided written informed consent.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | FOLFOX-4+P/XELOX+P | FOLFOX-4+BV/XELOX+BV
Number analyzed (Participants) | 701 | 699
days | 241.0 [227 to 254] | 316.0 [294 to 338]
Statistical Analysis 1: Comparison: FOLFOX-4+P/XELOX+P vs FOLFOX-4+BV/XELOX+BV; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.0001, Log Rank; Hazard Ratio (HR) = 0.63, 97.5% CI 2-sided [0.52 to 0.75]

6. Secondary Outcome: PFS by General Approach, Participants With Curative Surgery Not Censored: Non-inferiority of XELOX Versus FOLFOX-4
Description: PFS is defined as the time from randomization to disease progression (PD) or death due to any cause. Participants who underwent curative surgery after experiencing a sufficient shrinkage of their tumor were not censored at the date of surgery, but any relapse, new occurrence of colorectal cancer, or death was considered as an event. Non-inferiority analysis that followed the general approach took into account all tumor assessments obtained during the primary study treatment phase, the post-study treatment phase and those obtained during the follow-up phase. Non-inferiority of the XELOX-containing arms was compared with the FOLFOX-4-containing arms.
Time Frame: Baseline until disease progression or death, approximately 2 years 6 months
Population: EPP excluded participants from the ITT who had violated major protocol inclusion or exclusion criteria or participants who were randomized and did not receive at least one dose of capecitabine, 5-FU, oxaliplatin, or bevacizumab/placebo.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | FOLFOX-4/FOLFOX-4+P/FOLFOX-4+BV | XELOX/XELOX+P/XELOX+BV
Number analyzed (Participants) | 937 | 967
days | 260.0 [247 to 270] | 244.0 [230 to 255]
Statistical Analysis 1: Comparison: FOLFOX-4/FOLFOX-4+P/FOLFOX-4+BV vs XELOX/XELOX+P/XELOX+BV; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Hazard Ratio (HR) = 1.03, 97.5% CI 2-sided [0.92 to 1.15]

7. Secondary Outcome: PFS by General Approach, Participants With Curative Surgery Not Censored: Superiority of Chemotherapy Plus BV Over Chemotherapy Alone
Description: PFS is defined as the time from randomization to disease progression (PD) or death due to any cause. Participants who underwent curative surgery after experiencing a sufficient shrinkage of their tumor were not censored at the date of surgery, but any relapse, new occurrence of colorectal cancer, or death was considered as an event. Superiority analysis that followed the general approach took into account all tumor assessments obtained during the primary study treatment phase, the post-study treatment phase and those obtained during the follow-up phase. Superiority of the BV-containing arms was compared with the chemotherapy alone arms.
Time Frame: Baseline until disease progression or death, approximately 2 years 6 months
Population: The ITT population included all randomized participants who provided written informed consent.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | FOLFOX-4+P/XELOX+P | FOLFOX-4+BV/XELOX+BV
Number analyzed (Participants) | 701 | 699
days | 245.0 [230 to 258] | 287.0 [276 to 300]
Statistical Analysis 1: Comparison: FOLFOX-4+P/XELOX+P vs FOLFOX-4+BV/XELOX+BV; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.0015, Log Rank; Hazard Ratio (HR) = 0.83, 97.5% CI 2-sided [0.72 to 0.95]

8. Secondary Outcome: Overall Survival: Non-inferiority of XELOX Versus FOLFOX-4
Description: Overall survival was defined as the time from the date of randomization to the date of death. Participants who were not reported to have died at the time of the clinical cut-off date for the analysis were censored using the date they were last known to be alive. Non-inferiority of the XELOX-containing arms was compared with the FOLFOX-4-containing arms.
Time Frame: Baseline until disease progression or death, approximately 2 years 6 months
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | FOLFOX-4/FOLFOX-4+P/FOLFOX-4+BV | XELOX/XELOX+P/XELOX+BV
Number analyzed (Participants) | 937 | 967
days | 549.0 [528 to 576] | 577.0 [535 to 615]
Statistical Analysis 1: Comparison: FOLFOX-4/FOLFOX-4+P/FOLFOX-4+BV vs XELOX/XELOX+P/XELOX+BV; [analysis description as in outcome 4, analysis 1]; Test type: Non-Inferiority or Equivalence — This study was not powered for testing non-inferiority of XELOX vs FOLFOX-4 with respect to overall survival and no margin could be derived following the effect retention concept. The same margins used for the PFS analysis [Non-inferiority was demonstrated if the upper limit of the 2-sided 97.5% confidence interval (CI) for the hazard ratio (HR) was less than the predefined limit of 1.23 (the non-inferiority margin)] were therefore applied to OS as well; Hazard Ratio (HR) = 0.97, 97.5% CI 2-sided [0.84 to 1.14]

9. Secondary Outcome: Overall Survival: Superiority of Chemotherapy Plus BV Over Chemotherapy Alone
Description: Overall survival was defined as the time from the date of randomization to the date of death. Participants who were not reported to have died at the time of the clinical cut-off date for the analysis were censored using the date they were last known to be alive. Superiority of the BV-containing arms was compared with the chemotherapy alone arms.
Time Frame: Baseline until disease progression or death, approximately 2 years 6 months
Population: The ITT population included all randomized participants who provided written informed consent.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | FOLFOX-4+P/XELOX+P | FOLFOX-4+BV/XELOX+BV
Number analyzed (Participants) | 701 | 699
days | 574.0 [537 to 592] | 551.0 [528 to 635]
Statistical Analysis 1: Comparison: FOLFOX-4+P/XELOX+P vs FOLFOX-4+BV/XELOX+BV; Testing for superiority was based on the stratified log-rank test and used a two-sided significance level of 2.5%.The hazard ratio (HR) of bevacizumab in combination with chemotherapy versus chemotherapy alone [HR(FOLFOX-4+P/XELOX+P)/(FOLFOX-4+BV/XELOX+BV)] was presented together with the 97.5% confidence interval; Test type: Superiority or Other; p = 0.1921, Log Rank; Hazard Ratio (HR) = 0.89, 97.5% CI 2-sided [0.72 to 1.09]

10. Primary Outcome: PFS as Assessed by the Investigator According to Response Evaluation Criteria in Solid Tumors (RECIST) by General Approach (Participants With Curative Surgery Censored) - Superiority of Chemotherapy Plus BV Over Chemotherapy Alone
Description: PFS was defined as the time from randomization to progressive disease or death. Participants with neither disease progression nor death were censored at the last date of the last tumor assessment that confirmed that their disease had not progressed. Participants with no tumor assessments after baseline who were alive at the time of clinical cutoff were censored at the date of randomization. Participants who underwent surgical resection with curative intent without prior progression were censored at the date of surgery. PFS was based on tumor assessments made by the investigators according to the RECIST criteria. Superiority analysis that followed the general approach took into account all tumor assessments obtained during the primary study treatment phase, the post-study treatment phase and those obtained during the follow-up phase. Superiority of the BV-containing arms was compared with the chemotherapy alone arms.
Time Frame: Baseline until disease progression or death, approximately 2 years 6 months
Population: The ITT population included all randomized participants who provided written informed consent.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | FOLFOX-4+P/XELOX+P | FOLFOX-4+BV/XELOX+BV
Number analyzed (Participants) | 701 | 699
days | 244.0 [230 to 257] | 285.0 [271 to 297]
Statistical Analysis 1: Comparison: FOLFOX-4+P/XELOX+P vs FOLFOX-4+BV/XELOX+BV; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.0023, Log Rank; Hazard Ratio (HR) = 0.83, 97.5% CI 2-sided [0.72 to 0.95]

11. Secondary Outcome: Best Overall Response (BOR) as Assessed by the Investigator According to Response Evaluation Criteria in Solid Tumors (RECIST): Non-inferiority of XELOX Versus FOLFOX-4
Description: According to the RECIST criteria, BOR in an individual participant was defined as the best response recorded from the start of the treatment until disease progression or recurrence. Only tumor assessments as assessed by the investigator and made up to and including 28 days after last intake of study medication in the primary study treatment phase not later than date of first curative surgery were included in these analyses. Responders were defined as the percentage of participants with a confirmed best overall response of complete response (CR) or partial response (PR). Non-inferiority of the XELOX-containing arms was compared with the FOLFOX-4-containing arms.
Time Frame: From baseline until disease progression/recurrence, approximately 2 years 6 months
Population: as for outcome 2
Measure: Number; unit: Percentage of responders
Arm/Group | FOLFOX-4/FOLFOX-4+P/FOLFOX-4+BV | XELOX/XELOX+P/XELOX+BV
Number analyzed (Participants) | 937 | 967
Percentage of responders | 49.4 | 46.4
Statistical Analysis 1: Comparison: FOLFOX-4/FOLFOX-4+P/FOLFOX-4+BV vs XELOX/XELOX+P/XELOX+BV; Non-inferiority of XELOX with/without bevacizumab to FOLFOX-4 with/without bevacizumab was tested by the pair of hypotheses - H0: OR(XELOX/XELOX+P/XELOX+BV)/(FOLFOX-4/FOLFOX-4+P/FOLFOX-4+BV) </= 0.66 versus H1: OR(XELOX/XELOX+P/XELOX+BV)/(FOLFOX-4/FOLFOX-4+P/FOLFOX-4+BV) > 0.66, where OR denotes Odds ratio; Test type: Non-Inferiority or Equivalence — The analysis was based on the two-sided 97.5% confidence interval for OR(XELOX/XELOX+P/XELOX+BV)/(FOLFOX-4/FOLFOX-4+P/FOLFOX-4+BV). Non-inferiority of XELOX with/without bevacizumab to FOLFOX-4 with/without bevacizumab was concluded if the lower limit of this confidence interval is above 0.66; Odds Ratio (OR) = 0.89, 97.5% CI 2-sided [0.72 to 1.09]

12. Secondary Outcome: Best Overall Response (BOR) as Assessed by the Investigator According to RECIST: Superiority of Chemotherapy Plus BV Over Chemotherapy Alone
Description: According to the RECIST criteria, BOR in an individual participant was defined as the best response recorded from the start of the treatment until disease progression or recurrence. Only tumor assessments as assessed by the investigator and made up to and including 28 days after last intake of study medication in the primary study treatment phase not later than date of first curative surgery were included in these analyses. Responders were defined as the percentage of participants with a confirmed best overall response of complete response (CR) or partial response (PR). Superiority of the BV-containing arms was compared with the chemotherapy alone arms.
Time Frame: From baseline until disease progression/recurrence, approximately 2 years 6 months
Population: The ITT population included all randomized participants who provided written informed consent.
Measure: Number; unit: Percentage of responders
Arm/Group | FOLFOX-4+P/XELOX+P | FOLFOX-4+BV/XELOX+BV
Number analyzed (Participants) | 701 | 699
Percentage of responders | 49.2 | 46.5
Statistical Analysis 1: Comparison: FOLFOX-4+P/XELOX+P vs FOLFOX-4+BV/XELOX+BV; Superiority of adding bevacizumab to chemotherapy was tested as follows - H0: OR(FOLFOX-4+BV/XELOX+BV)/(FOLFOX-4+P/XELOX+P) </= 1.0 versus H1: OR(FOLFOX-4+BV/XELOX+BV)/(FOLFOX-4+P/XELOX+P) > 1.0. The test used a two-sided significance level of 2.5%; Test type: Superiority or Other; p = 0.3091, Chi-squared; Odds Ratio (OR) = 0.90, 97.5% CI 2-sided [0.71 to 1.14]

13. Secondary Outcome: BOR as Assessed by the IRC According to RECIST: Non-inferiority of XELOX Versus FOLFOX-4
Description: According to the RECIST criteria, the BOR in an individual participant was the best response recorded from the start of the treatment until disease progression/recurrence (taking the smallest measurements recorded since the baseline assessment as a reference for PD). The BOR as assessed by the IRC was determined based on tumor assessments that were made up to and including 28 days after last intake of study medication in the primary study treatment phase. Responders were defined as the percentage of participants with a complete response (CR) or partial response (PR). Non-inferiority of the XELOX-containing arms was compared with the FOLFOX-4-containing arms.
Time Frame: From baseline until disease progression/recurrence, approximately 2 years 6 months
Population: as for outcome 2
Measure: Number; unit: Percentage of responders
Arm/Group | FOLFOX-4/FOLFOX-4+P/FOLFOX-4+BV | XELOX/XELOX+P/XELOX+BV
Number analyzed (Participants) | 937 | 967
Percentage of responders | 38.6 | 37.1
Statistical Analysis 1: Comparison: FOLFOX-4/FOLFOX-4+P/FOLFOX-4+BV vs XELOX/XELOX+P/XELOX+BV; Non-inferiority of XELOX with/without bevacizumab to FOLFOX-4 with/without bevacizumab was tested by the pair of hypotheses - H0: OR(XELOX/XELOX+P/XELOX+BV)/(FOLFOX-4/FOLFOX-4+P/FOLFOX-4+BV) </= 0.66 versus H1: OR(XELOX/XELOX+P/XELOX+BV)/(FOLFOX-4/FOLFOX-4+P/FOLFOX-4+BV) > 0.66; Test type: Non-Inferiority or Equivalence — The analysis was based on the two-sided 97.5% confidence interval for OR(XELOX/XELOX+P/XELOX+BV)/(FOLFOX-4/FOLFOX-4+P/FOLFOX-4+BV). Non-inferiority of XELOX with/without bevacizumab to FOLFOX-4 with/without bevacizumab shall be concluded if the lower limit of this confidence interval is above 0.66; Odds Ratio (OR) = 0.94, 97.5% CI 2-sided [0.76 to 1.16]

14. Secondary Outcome: BOR as Assessed by the IRC According to RECIST: Superiority of Chemotherapy Plus BV Over Chemotherapy Alone
Description: According to the RECIST criteria, the BOR in an individual participant was the best response recorded from the start of the treatment until disease progression/recurrence (taking the smallest measurements recorded since the baseline assessment as a reference for PD). The BOR as assessed by the IRC was determined based on tumor assessments that were made up to and including 28 days after last intake of study medication in the primary study treatment phase. Responders were defined as the percentage of participants with a complete response (CR) or partial response (PR). Superiority of the BV-containing arms was compared with the chemotherapy alone arms.
Time Frame: From baseline until disease progression/recurrence, approximately 2 years 6 months
Population: The ITT population included all randomized participants who provided written informed consent.
Measure: Number; unit: Percentage of responders
Arm/Group | FOLFOX-4+P/XELOX+P | FOLFOX-4+BV/XELOX+BV
Number analyzed (Participants) | 701 | 699
Percentage of responders | 37.5 | 37.5
Statistical Analysis 1: Comparison: FOLFOX-4+P/XELOX+P vs FOLFOX-4+BV/XELOX+BV; Superiority of adding bevacizumab to chemotherapy was tested as follows - H0: OR(FOLFOX-4+BV/XELOX+BV)/(FOLFOX 4+P/XELOX+P) </= 1.0 versus H1: OR(FOLFOX-4+BV/XELOX+BV)/(FOLFOX-4+P/XELOX+P) > 1.0. The test used a two-sided significance level of 2.5%; Test type: Superiority or Other; p = 0.9887, Chi-squared; Odds Ratio (OR) = 1.00, 97.5% CI 2-sided [0.78 to 1.28]

15. Secondary Outcome: Time to Treatment Failure (TTF) as Assessed by the Investigator According to RECIST: Non-inferiority of XELOX Versus FOLFOX-4
Description: Time to treatment failure was defined as the time from the date of randomization to the date of discontinuation of the primary study treatment phase due to adverse event/intercurrent illness, insufficient therapeutic response, death, failure to return, refusing treatment/being unwilling to cooperate, or withdrawing consent; discontinuation of the post study treatment phase due to adverse event, progressive disease, death, participant refusal/administrative reasons, or withdrawing consent; documented disease progression; or death due to any cause, whichever occurred first. The general approach took into account all tumor assessments obtained during the primary study treatment phase, the post-study treatment phase and those obtained during the follow-up phase.The on-treatment approach included only tumor assessments and deaths that occurred no later than 28 days after the last confirmed intake of any study medication in the primary study treatment phase only.
Time Frame: From baseline until disease progression/recurrence, approximately 2 years 6 months
Population: The safety population included all participants who were randomized and received at least one dose of capecitabine, 5-FU, oxaliplatin, or bevacizumab/placebo.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | FOLFOX-4/FOLFOX-4+P/FOLFOX-4+BV | XELOX/XELOX+P/XELOX+BV
Number analyzed (Participants) | 990 | 1008
days
  General Approach | 191.0 [183 to 202] | 179.0 [171 to 187]
  On-treatment Approach | 190.0 [182 to 200] | 176.0 [170 to 185]
Statistical Analysis 1: Comparison: FOLFOX-4/FOLFOX-4+P/FOLFOX-4+BV vs XELOX/XELOX+P/XELOX+BV; General approach: HRs and 97.5% confidence interval were reported for treatment arm A (XELOX/XELOX+P/XELOX+BV) versus treatment arm B (FOLFOX-4/FOLFOX-4+P/FOLFOX-4+BV); Test type: Non-Inferiority or Equivalence — No formal statistical testing was done; Hazard Ratio (HR) = 1.08, 97.5% CI 2-sided [0.97 to 1.20]
Statistical Analysis 2: Comparison: FOLFOX-4/FOLFOX-4+P/FOLFOX-4+BV vs XELOX/XELOX+P/XELOX+BV; On-treatment Approach: HRs and 97.5% confidence interval were reported for treatment arm A (XELOX/XELOX+P/XELOX+BV) versus treatment arm B (FOLFOX-4/FOLFOX-4+P/FOLFOX-4+BV); Test type: Non-Inferiority or Equivalence — Fewer events were expected in analyses using the on-treatment approach than in the analyses using the general approach, thus leading to reduced power.Therefore, no formal statistical testing was performed; Hazard Ratio (HR) = 1.10, 97.5% CI 2-sided [0.98 to 1.23]

16. Secondary Outcome: Time to Treatment Failure as Assessed by the Investigator According to RECIST: Superiority of Chemotherapy Plus BV Over Chemotherapy Alone
Description: Time to treatment failure was defined as the time from the date of randomization to the date of discontinuation of the primary study treatment phase due to adverse event/intercurrent illness, insufficient therapeutic response, death, failure to return, refusing treatment/being unwilling to cooperate, or withdrawing consent; discontinuation of the post study treatment phase due to adverse event, progressive disease, death, participant refusal/administrative reasons, or withdrawing consent; documented disease progression; or death due to any cause, whichever occurred first. The general approach included all tumor assessments or deaths that occurred during the primary study treatment phase, the post-study treatment phase, or the follow-up phase. The on-treatment approach included only tumor assessments and deaths that occurred no later than 28 days after the last confirmed intake of any study medication in the primary study treatment phase only.
Time Frame: From baseline until disease progression/recurrence, approximately 2 years 6 months
Population: as for outcome 15
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | FOLFOX-4+P/XELOX+P | FOLFOX-4+BV/XELOX+BV
Number analyzed (Participants) | 675 | 694
days
  General Approach | 183.0 [176 to 198] | 209.0 [199 to 220]
  On-treatment Approach | 182.0 [175 to 196] | 208.0 [198 to 220]
Statistical Analysis 1: Comparison: FOLFOX-4+P/XELOX+P vs FOLFOX-4+BV/XELOX+BV; General approach: Testing for superiority was based on the stratified log-rank test and used a two-sided significance level of 2.5%.The hazard ratio (HR) of bevacizumab in combination with chemotherapy versus chemotherapy alone [HR(FOLFOX-4+P/XELOX+P)/(FOLFOX-4+BV/XELOX+BV)] was presented; Test type: Superiority or Other; p = 0.0030, Log Rank; Hazard Ratio (HR) = 0.84, 97.5% CI 2-sided [0.74 to 0.96]
Statistical Analysis 2: Comparison: FOLFOX-4+P/XELOX+P vs FOLFOX-4+BV/XELOX+BV; On treatment approach: Testing for superiority was based on the stratified log-rank test and used a two-sided significance level of 2.5%.The hazard ratio (HR) of bevacizumab in combination with chemotherapy versus chemotherapy alone [HR(FOLFOX-4+P/XELOX+P)/(FOLFOX-4+BV/XELOX+BV)] was presented; Test type: Superiority or Other; p = 0.0004, Log Rank; Hazard Ratio (HR) = 0.81, 97.5% CI 2-sided [0.70 to 0.92]

17. Secondary Outcome: Time to Response as Assessed by the Investigator According to RECIST: Non-inferiority of XELOX Versus FOLFOX-4
Description: For participants whose BOR was CR or PR, time to response was measured as the time from randomization to the first time when the measurement criteria for CR or PR (whichever status was recorded first) was met. It was based on tumor assessments made by the investigators according to the RECIST criteria. Results were reported as the number of participants achieving a response in 8 time categories from Week 1 to Week 54. Non-inferiority of the XELOX-containing arms was compared with the FOLFOX-4-containing arms.
Time Frame: Week 1 to Week 54
Population: as for outcome 2
Measure: Number; unit: Participants
Arm/Group | FOLFOX-4/FOLFOX-4+P/FOLFOX-4+BV | XELOX/XELOX+P/XELOX+BV
Number analyzed (Participants) | 937 | 967
Participants
  Week 1-6 | 67 | 93
  Week 7-12 | 190 | 191
  Week 13-18 | 155 | 110
  Week 19-24 | 25 | 38
  Week 25-30 | 14 | 13
  Week 31-36 | 7 | 3
  Week 37-42 | 3 | 1
  Week 49-54 | 2 | 0

18. Secondary Outcome: Time to Response as Assessed by the Investigator According to RECIST: Superiority of Chemotherapy Plus BV Over Chemotherapy Alone
Description: For participants whose BOR was CR or PR, time to response was measured as the time from randomization to the first time when the measurement criteria for CR or PR (whichever status was recorded first) was met. It was based on tumor assessments made by the investigators according to the RECIST criteria. Results were reported as the number of participants achieving a response in 8 time categories from Week 1 to Week 54. Superiority of the BV-containing arms was compared with the chemotherapy alone arms.
Time Frame: Week 1 to Week 54
Population: The ITT population included all randomized participants who provided written informed consent.
Measure: Number; unit: Participants
Arm/Group | FOLFOX-4+P/XELOX+P | XELOX/XELOX+P/XELOX+BV
Number analyzed (Participants) | 701 | 699
Participants
  Week 1-6 | 58 | 48
  Week 7-12 | 146 | 138
  Week 13-18 | 105 | 87
  Week 19-24 | 26 | 29
  Week 25-30 | 7 | 12
  Week 31-36 | 2 | 8
  Week 37-42 | 1 | 2
  Week 49-54 | 0 | 1

19. Secondary Outcome: Duration of Overall Response as Assessed by the Investigator According to RECIST: Non-inferiority of XELOX Versus FOLFOX-4
Description: Duration of overall response was measured from the time that measurement criteria were first met for CR or PR (whichever status was recorded first) until the first date when progressive disease or death was documented. It was based on tumor assessments made by the investigators according to the RECIST criteria. Participants who neither progressed nor died were censored at the date of the last tumor assessment. Participants undergoing surgical resection with curative intent were censored at the date of surgery. Non-inferiority of the XELOX-containing arms was compared with the FOLFOX-4-containing arms.
Time Frame: From baseline until disease progression/recurrence, approximately 2 years 6 months
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | FOLFOX-4/FOLFOX-4+P/FOLFOX-4+BV | XELOX/XELOX+P/XELOX+BV
Number analyzed (Participants) | 937 | 967
days | 239.0 [225 to 256] | 226.0 [211 to 246]
Statistical Analysis 1: Comparison: FOLFOX-4/FOLFOX-4+P/FOLFOX-4+BV vs XELOX/XELOX+P/XELOX+BV; [analysis description as in outcome 4, analysis 1]; Test type: Non-Inferiority or Equivalence — No formal statistical testing was performed for duration of overall response; Hazard Ratio (HR) = 1.02, 97.5% CI 2-sided [0.86 to 1.22]

20. Secondary Outcome: Duration of Overall Response as Assessed by the Investigator According to RECIST: Superiority Analysis of Chemotherapy Plus Bevacizumab Versus Chemotherapy Alone
Description: Duration of overall response was measured from the time that measurement criteria were first met for CR or PR (whichever status was recorded first) until the first date when progressive disease or death was documented. It was based on tumor assessments made by the investigators according to the RECIST criteria. Participants who neither progressed nor died were censored at the date of the last tumor assessment. Participants undergoing surgical resection with curative intent were censored at the date of surgery. Superiority of the BV-containing arms was compared with the chemotherapy alone arms.
Time Frame: From baseline until disease progression/recurrence, approximately 2 years 6 months
Population: The ITT population included all randomized participants who provided written informed consent.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | FOLFOX-4+P/XELOX+P | FOLFOX-4+BV/XELOX+BV
Number analyzed (Participants) | 701 | 699
days | 225.0 [217 to 240] | 257.0 [241 to 278]
Statistical Analysis 1: Comparison: FOLFOX-4+P/XELOX+P vs FOLFOX-4+BV/XELOX+BV; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.0307, Log Rank; Hazard Ratio (HR) = 0.82, 97.5% CI 2-sided [0.66 to 1.01]

21. Secondary Outcome: Duration of Complete Response as Assessed by the Investigator According to RECIST: Non-inferiority of XELOX Versus FOLFOX-4
Description: For complete responders, the duration of complete response was measured from the time measurement criteria were first met for complete response until the date that progressive disease (or death) was documented. Non-inferiority of the XELOX-containing arms was compared with the FOLFOX-4-containing arms.
Time Frame: From baseline until disease progression/recurrence, approximately 2 years 6 months
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | FOLFOX-4/FOLFOX-4+P/FOLFOX-4+BV | XELOX/XELOX+P/XELOX+BV
Number analyzed (Participants) | 937 | 967
days | 347.0 [196 to 403] | 589.0 [270 to NA] — The estimate is Not Available due to insufficient follow-up time to estimate the missing parameter.
Statistical Analysis 1: Comparison: FOLFOX-4/FOLFOX-4+P/FOLFOX-4+BV vs XELOX/XELOX+P/XELOX+BV; [analysis description as in outcome 4, analysis 1]; Test type: Non-Inferiority or Equivalence — No formal statistical testing was done; Hazard Ratio (HR) = 0.35, 97.5% CI 2-sided [0.09 to 1.39]

22. Secondary Outcome: Duration of Complete Response as Assessed by the Investigator According to RECIST: Superiority of Chemotherapy Plus BV Over Chemotherapy Alone
Description: For complete responders, the duration of complete response was measured from the time measurement criteria were first met for complete response until the date that progressive disease (or death) was documented. Superiority of the BV-containing arms was compared with the chemotherapy alone arms.
Time Frame: From baseline until disease progression/recurrence, approximately 2 years 6 months
Population: The ITT population included all randomized participants who provided written informed consent.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | FOLFOX-4+P/XELOX+P | FOLFOX-4+BV/XELOX+BV
Number analyzed (Participants) | 701 | 699
days | 403.0 [228 to NA] — The estimate is Not Available due to insufficient follow-up time to estimate the missing parameter. | 386.0 [133 to 386]
Statistical Analysis 1: Comparison: FOLFOX-4+P/XELOX+P vs FOLFOX-4+BV/XELOX+BV; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.8207, Log Rank; Hazard Ratio (HR) = 1.20, 97.5% CI 2-sided [0.20 to 7.05]

ADVERSE EVENTS:
Time Frame: Approximately 2 years 6 months
Description: Serious adverse events (SAEs) and non-serious adverse events were reported for members of the safety population, which included all participants were randomized and received at least one dose of capecitabine, 5-FU, oxaliplatin, or bevacizumab/placebo.
Arm/Group | Xelox | Folfox-4 | Xelox+P | Folfox-4+P | Xelox+BV | Folfox-4+BV
Serious Adverse Events (participants affected / at risk) | 117/316 | 120/313 | 121/339 | 128/336 | 131/353 | 146/341
Other Adverse Events (participants affected / at risk) | 310/316 | 310/313 | 330/339 | 331/336 | 348/353 | 335/341
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Xelox (N=316) | Folfox-4 (N=313) | Xelox+P (N=339) | Folfox-4+P (N=336) | Xelox+BV (N=353) | Folfox-4+BV (N=341)
Diarrhoea (Gastrointestinal disorders) | 27 | 13 | 25 | 7 | 26 | 8
Vomiting (Gastrointestinal disorders) | 7 | 7 | 16 | 2 | 14 | 7
Abdominal pain (Gastrointestinal disorders) | 4 | 7 | 7 | 6 | 5 | 7
Intestinal obstruction (Gastrointestinal disorders) | 4 | 6 | 6 | 9 | 4 | 6
Small intestinal obstruction (Gastrointestinal disorders) | 5 | 3 | 3 | 2 | 4 | 7
Nausea (Gastrointestinal disorders) | 1 | 6 | 4 | 0 | 5 | 2
Constipation (Gastrointestinal disorders) | 1 | 5 | 1 | 3 | 3 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 2 | 3 | 1 | 0 | 3
Ascites (Gastrointestinal disorders) | 3 | 0 | 1 | 1 | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 2 | 2 | 0 | 4 | 1
Stomatitis all (Gastrointestinal disorders) | 2 | 0 | 0 | 1 | 1 | 2
Enteritis (Gastrointestinal disorders) | 3 | 0 | 1 | 1 | 0 | 0
Intestinal perforation (Gastrointestinal disorders) | 1 | 1 | 1 | 0 | 2 | 1
Abdominal pain upper (Gastrointestinal disorders) | 1 | 1 | 1 | 1 | 0 | 1
Ileus (Gastrointestinal disorders) | 0 | 1 | 2 | 0 | 2 | 0
Colitis (Gastrointestinal disorders) | 1 | 0 | 0 | 2 | 1 | 0
Haematemesis (Gastrointestinal disorders) | 0 | 0 | 1 | 2 | 0 | 0
Large intestinal obstruction (Gastrointestinal disorders) | 1 | 1 | 1 | 0 | 1 | 0
Mechanical ileus (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0 | 1
Gastrointestinal toxicity (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 0 | 0
Intestinal functional disorder (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Melaena (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0 | 0
Abdominal adhesions (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Caecitis (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 0 | 0
Enterocolitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 1
Enterovesical fistula (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 0
Gastrointestinal disorder (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2 | 0
Gastrointestinal hypomotility (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 1
Gastrointestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 0
Ileus paralytic (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 0
Intestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Pericoronitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Peritonitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 1
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Anal fissure (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Anal stenosis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Colonic obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Crohn's disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Duodenal ulcer (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Enterocolonic fistula (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Faecaloma (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Gastrointestinal necrosis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Gastrointestinal perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Inguinal hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Intestinal ischemia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Oesophagitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Proctalgia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Rectal perforation (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Subileus (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Toxic dilatation of intestine (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Central line infection (Infections and infestations) | 1 | 4 | 1 | 9 | 0 | 4
Pneumonia (Infections and infestations) | 2 | 5 | 4 | 3 | 4 | 3
Infection (Infections and infestations) | 0 | 1 | 1 | 4 | 0 | 5
Sepsis (Infections and infestations) | 4 | 4 | 1 | 2 | 4 | 4
Urinary tract infection (Infections and infestations) | 1 | 1 | 3 | 5 | 1 | 1
Septic shock (Infections and infestations) | 1 | 2 | 1 | 1 | 2 | 2
Cellulitis (Infections and infestations) | 2 | 1 | 2 | 0 | 0 | 2
Catheter site infection (Infections and infestations) | 0 | 2 | 0 | 2 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 1 | 1 | 1 | 1 | 0 | 0
Neutropenic sepsis (Infections and infestations) | 0 | 2 | 0 | 1 | 0 | 2
Diverticulitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Abdominal abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 2
Bacteraemia (Infections and infestations) | 0 | 0 | 1 | 0 | 2 | 0
Respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 2
Bacterial sepsis (Infections and infestations) | 0 | 1 | 0 | 1 | 0 | 0
Clostridium difficile colitis (Infections and infestations) | 1 | 0 | 1 | 0 | 0 | 0
Postoperative wound infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Abdominal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Abdominal wall infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 2
Diarrhoea infectious (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 1 | 0 | 1 | 0 | 0 | 0
Gastrointestinal infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Hepatitis B (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Pneumonia pneumococcal (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Pyelonephritis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Urosepsis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Viral pharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Abdominal wall abscess (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Acinetobacter bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Anal fistula infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Bacterial infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Bronchitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Bronchopneumonia (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Catheter related infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Catheter sepsis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Fungaemia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Neutropenic infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Peritoneal infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Pseudomonas infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Pyonephrosis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Rectal abscess (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Staphylococcal infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Staphylococcal sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 16 | 16 | 6 | 16 | 7 | 15
Asthenia (General disorders) | 1 | 1 | 2 | 0 | 1 | 0
Chest pain (General disorders) | 2 | 1 | 1 | 0 | 1 | 2
Catheter related complication (General disorders) | 1 | 2 | 1 | 2 | 0 | 2
Fatigue (General disorders) | 0 | 1 | 0 | 0 | 1 | 1
General physical health deterioration (General disorders) | 2 | 0 | 1 | 1 | 1 | 1
Oedema peripheral (General disorders) | 0 | 2 | 0 | 1 | 0 | 0
Multi-organ failure (General disorders) | 0 | 1 | 0 | 0 | 2 | 2
Performance status decreased (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
Extravasation (General disorders) | 0 | 0 | 0 | 0 | 1 | 1
Non-cardiac chest pain (General disorders) | 1 | 0 | 1 | 0 | 0 | 0
Pain (General disorders) | 0 | 0 | 1 | 1 | 0 | 0
Infusion related reaction (General disorders) | 0 | 0 | 0 | 1 | 0 | 1
Sudden death (General disorders) | 0 | 0 | 0 | 0 | 2 | 0
Wound necrosis (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
Chills (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Impaired healing (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
Oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 3 | 14 | 1 | 15 | 2 | 14
Neutropenia (Blood and lymphatic system disorders) | 2 | 9 | 1 | 6 | 0 | 5
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 2 | 2 | 1 | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 1 | 2 | 1 | 3 | 0 | 1
Blood disorder (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Coagulopathy (Blood and lymphatic system disorders) | 1 | 1 | 0 | 0 | 1 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 2
Agranulocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Haemolytic anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Pancytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Thrombotic thrombocytopenic purpura (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 9 | 3 | 3 | 5 | 9 | 8
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2 | 3 | 4 | 3
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 1 | 3 | 2
Dysaesthesia pharynx (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 4 | 0 | 2 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 1 | 1 | 3
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 1 | 1
Alveolitis fibrosing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 1 | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 1 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Laryngospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 4 | 9 | 10 | 2 | 10 | 4
Hypokalaemia' (Metabolism and nutrition disorders) | 2 | 0 | 1 | 1 | 2 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 2 | 0 | 2 | 1
Anorexia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 1 | 0
Hypernatraemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0 | 0 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 1 | 0
Malnutrition (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0
Cachexia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0
Hypovolaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 6 | 6 | 1 | 7 | 7 | 6
Thrombosis (Vascular disorders) | 2 | 0 | 1 | 2 | 2 | 1
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 2 | 1
Jugular vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 2 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 1 | 1 | 0 | 1
Thrombophlebitis (Vascular disorders) | 0 | 0 | 0 | 1 | 1 | 1
Embolism (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 2
Peripheral ischaemia (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 1
Hypertensive crisis (Vascular disorders) | 0 | 0 | 0 | 0 | 2 | 0
Pelvic venous thrombosis (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 1
Venous thrombosis limb (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0
Circulatory collapse (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0
Embolism venous (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0
Haematoma (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0
Haemorrhage (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0
Hypovolaemic shock (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0
Poor venous access (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0
Shock (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1
Shock haemorrhagic (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0
Subclavian vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0
Venous thrombosis (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 0 | 1 | 4 | 2
Myocardial infarction (Cardiac disorders) | 0 | 3 | 0 | 0 | 0 | 3
Pericardial effusion (Cardiac disorders) | 2 | 0 | 0 | 0 | 0 | 0
Cardiac arrest (Cardiac disorders) | 0 | 1 | 0 | 1 | 2 | 0
Angina pectoris (Cardiac disorders) | 1 | 1 | 0 | 0 | 0 | 1
Cardiomyopathy (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0
Myocardial ischaemia (Cardiac disorders) | 0 | 0 | 0 | 0 | 2 | 1
Arrhythmia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 1
Acute left ventricular failure (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0
Atrial thrombosis (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0
Bradycardia (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1
Cardio-respiratory arrest (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1
Cardiogenic shock (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0
Cardiopulmonary failure (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0
Sick sinus syndrome (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1
Ventricular fibrillation (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 2 | 0 | 0 | 0 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Convulsion (Nervous system disorders) | 1 | 1 | 0 | 1 | 1 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 1 | 1 | 1
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 0 | 1 | 1 | 1
Headache (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 0 | 1 | 1 | 1 | 0
Cerebral infarction (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Coordination abnormal (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Dementia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Loss of consciousness (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 1
Neuralgia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Spinal cord compression (Nervous system disorders) | 1 | 0 | 1 | 0 | 0 | 0
Cerebral haemorrhage (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Cerebral ischaemia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Depressed level of consciousness (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Encephalophathy (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Hepatic encephalopathy (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0 | 1 | 0
Gastrointestinal stoma complication (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 2 | 0 | 0
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1 | 0 | 0
Stent occlussion (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Femur fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 1
Head injury (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0 | 0 | 0
Radius fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Device migration (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0
Failure to anastomose (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Hip fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0
Overdose (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Skull fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Tendon rupture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Ulna fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Vascular graft occlussion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Renal failure acute (Renal and urinary disorders) | 1 | 0 | 3 | 0 | 3 | 2
Renal failure (Renal and urinary disorders) | 1 | 0 | 1 | 1 | 2 | 0
Haematuria (Renal and urinary disorders) | 3 | 1 | 0 | 0 | 0 | 0
Hydronephrosis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0
Renal colic (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 1
Urinary bladder haemmorhage (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0
Urinary retention (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 1 | 0
Obstructive uropathy (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0
Renal impairment (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0
Renal tubular disorder (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0
Renal tubular necrosis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0
Ureteric obstruction (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0
Hepatic failure (Hepatobiliary disorders) | 1 | 0 | 0 | 1 | 1 | 0
Bile duct obstruction (Hepatobiliary disorders) | 1 | 1 | 0 | 2 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1
Portal vein thrombosis (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 1 | 1
Cholangitis (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 1 | 0 | 1 | 0 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0
Hepatitis (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0 | 0
Hepatitis Cholestatic (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 2 | 0 | 0 | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Muscle contracture (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 1
Shoulder pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Hypersensitivity (Immune system disorders) | 0 | 0 | 2 | 2 | 2 | 2
Drug hypersensitivity (Immune system disorders) | 0 | 0 | 2 | 3 | 0 | 0
Anaphylactic reaction (Immune system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Anaphylactic shock (Immune system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2 | 0 | 1 | 0
Tumor haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 1
Colon neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0
Gastric neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0
Metastases to ovary (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0
Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 1
Transaminases increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
International normalized ratio increased (Investigations) | 0 | 0 | 0 | 1 | 1 | 0
Blood bilirubin abnormal (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
Endoscopic retrograde cholangiopancreatography (Investigations) | 0 | 1 | 0 | 0 | 0 | 0
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Angioneurotic oedema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Skin toxicity (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Vascular purpura (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Confusional state (Psychiatric disorders) | 1 | 1 | 1 | 0 | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0 | 1
Retinal vascular thrombosis (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0
Amaurosis (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0
Catheter placement (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 0 | 1
Colostomy closure (Surgical and medical procedures) | 0 | 0 | 1 | 0 | 0 | 0
Ileostomy closure (Surgical and medical procedures) | 0 | 0 | 1 | 0 | 0 | 0
Vaginal fistula (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Xelox (N=316) | Folfox-4 (N=313) | Xelox+P (N=339) | Folfox-4+P (N=336) | Xelox+BV (N=353) | Folfox-4+BV (N=341)
Diarrhoea (Gastrointestinal disorders) | 207 | 186 | 208 | 197 | 210 | 218
Nausea (Gastrointestinal disorders) | 194 | 208 | 209 | 204 | 230 | 215
Vomiting (Gastrointestinal disorders) | 136 | 123 | 134 | 127 | 160 | 127
Stomatitis All (Gastrointestinal disorders) | 63 | 111 | 76 | 130 | 101 | 141
Constipation (Gastrointestinal disorders) | 73 | 78 | 77 | 99 | 68 | 101
Abdominal pain (Gastrointestinal disorders) | 81 | 76 | 86 | 89 | 85 | 81
Dyspepsia (Gastrointestinal disorders) | 30 | 53 | 41 | 35 | 30 | 40
Abdominal pain upper (Gastrointestinal disorders) | 25 | 27 | 28 | 43 | 32 | 34
Dry mouth (Gastrointestinal disorders) | 10 | 16 | 11 | 20 | 7 | 19
Paraesthesia (Nervous system disorders) | 116 | 117 | 126 | 127 | 133 | 135
Peripheral Sensory Neuropathy (Nervous system disorders) | 48 | 31 | 60 | 70 | 64 | 72
Neuropathy Peripheral (Nervous system disorders) | 64 | 70 | 64 | 60 | 70 | 61
Dysaesthesia (Nervous system disorders) | 37 | 38 | 43 | 50 | 46 | 42
Neuropathy (Nervous system disorders) | 42 | 33 | 51 | 51 | 50 | 48
Lethargy (Nervous system disorders) | 34 | 46 | 30 | 20 | 29 | 27
Headache (Nervous system disorders) | 41 | 34 | 36 | 50 | 53 | 62
Dysgeusia (Nervous system disorders) | 46 | 48 | 39 | 56 | 42 | 49
Hypoaesthesia (Nervous system disorders) | 32 | 29 | 20 | 14 | 16 | 15
Dizziness (Nervous system disorders) | 45 | 42 | 40 | 45 | 28 | 36
Neurotoxicity (Nervous system disorders) | 19 | 12 | 9 | 7 | 9 | 15
Fatigue (General disorders) | 132 | 152 | 118 | 140 | 133 | 135
Asthenia (General disorders) | 43 | 41 | 81 | 90 | 77 | 97
Pyrexia (General disorders) | 43 | 76 | 66 | 84 | 66 | 82
Temperature Intolerance (General disorders) | 21 | 29 | 31 | 18 | 31 | 22
Oedema Peripheral (General disorders) | 28 | 36 | 23 | 21 | 27 | 15
Chills (General disorders) | 10 | 18 | 16 | 23 | 12 | 20
Chest pain (General disorders) | 10 | 14 | 14 | 15 | 27 | 28
Neutropenia (Blood and lymphatic system disorders) | 88 | 172 | 90 | 198 | 70 | 187
Thrombocytopenia (Blood and lymphatic system disorders) | 85 | 70 | 61 | 78 | 48 | 44
Anaemia (Blood and lymphatic system disorders) | 50 | 37 | 41 | 40 | 31 | 38
Leukopenia (Blood and lymphatic system disorders) | 10 | 24 | 7 | 15 | 6 | 25
Palmar-Plantar Erythrodysaesthesia Syndrome (Skin and subcutaneous tissue disorders) | 95 | 30 | 103 | 36 | 138 | 46
Alopecia (Skin and subcutaneous tissue disorders) | 19 | 52 | 18 | 62 | 13 | 53
Rash (Skin and subcutaneous tissue disorders) | 14 | 32 | 31 | 34 | 25 | 40
Pruritus (Skin and subcutaneous tissue disorders) | 11 | 20 | 9 | 20 | 11 | 20
Dry skin (Skin and subcutaneous tissue disorders) | 15 | 17 | 21 | 15 | 26 | 17
Erythema (Skin and subcutaneous tissue disorders) | 11 | 18 | 13 | 12 | 11 | 14
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 22 | 41 | 24 | 62 | 38 | 107
Dysaesthesia pharynx (Respiratory, thoracic and mediastinal disorders) | 41 | 21 | 45 | 23 | 33 | 14
Cough (Respiratory, thoracic and mediastinal disorders) | 36 | 40 | 32 | 47 | 28 | 42
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 37 | 20 | 34 | 36 | 39 | 29
Hiccups (Respiratory, thoracic and mediastinal disorders) | 14 | 21 | 17 | 13 | 13 | 21
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 17 | 16 | 12 | 27 | 19 | 26
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 9 | 16 | 10 | 20 | 22 | 22
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 5 | 3 | 6 | 5 | 21 | 28
Anorexia (Metabolism and nutrition disorders) | 95 | 93 | 84 | 86 | 109 | 96
Hypokalaemia (Metabolism and nutrition disorders) | 35 | 32 | 31 | 21 | 26 | 21
Decreased appetite (Metabolism and nutrition disorders) | 16 | 15 | 14 | 10 | 9 | 18
Dehydration (Metabolism and nutrition disorders) | 28 | 16 | 17 | 11 | 20 | 11
Pain in extremity (Musculoskeletal and connective tissue disorders) | 43 | 20 | 35 | 26 | 43 | 34
Pain in jaw (Musculoskeletal and connective tissue disorders) | 23 | 16 | 13 | 16 | 15 | 12
Back pain (Musculoskeletal and connective tissue disorders) | 33 | 27 | 28 | 38 | 29 | 30
Muscle spasms (Musculoskeletal and connective tissue disorders) | 17 | 10 | 16 | 13 | 9 | 15
Arthralgia (Musculoskeletal and connective tissue disorders) | 13 | 16 | 12 | 24 | 21 | 20
Myalgia (Musculoskeletal and connective tissue disorders) | 9 | 9 | 18 | 14 | 11 | 10
Insomnia (Psychiatric disorders) | 33 | 44 | 31 | 46 | 30 | 40
Depression (Psychiatric disorders) | 20 | 13 | 23 | 14 | 14 | 10
Anxiety (Psychiatric disorders) | 14 | 16 | 17 | 14 | 16 | 7
Nasopharyngitis (Infections and infestations) | 9 | 18 | 27 | 36 | 26 | 39
Urinary tract infection (Infections and infestations) | 11 | 17 | 11 | 28 | 22 | 19
Upper respiratory tract infection (Infections and infestations) | 12 | 21 | 7 | 14 | 18 | 16
Hypertension (Vascular disorders) | 3 | 10 | 16 | 22 | 49 | 63
Flushing (Vascular disorders) | 7 | 22 | 4 | 7 | 9 | 8
Weight decreased (Investigations) | 27 | 27 | 35 | 25 | 45 | 32
Proteinuria (Renal and urinary disorders) | 1 | 0 | 10 | 21 | 14 | 22
Dysuria (Renal and urinary disorders) | 6 | 7 | 6 | 17 | 9 | 10
Lacrimation increased (Eye disorders) | 8 | 20 | 17 | 19 | 15 | 30
Hyperbilirubinaemia (Hepatobiliary disorders) | 10 | 4 | 18 | 6 | 11 | 3
Hypersensitivity (Immune system disorders) | 5 | 9 | 5 | 22 | 10 | 18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.